CLINICAL TRIAL: NCT02131532
Title: A Feasibility Study of a Brief Psychological Intervention for Post-stroke Fatigue
Brief Title: A Rehabilitation Therapy for Post-stroke Fatigue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSF-14/SS/0093
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2015-07

CONDITIONS: Stroke
Keywords: Post-stroke fatigue; Psychological intervention; Feasibility
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychological intervention (Experimental): This is a brief psychological intervention which targets patients' mood, their beliefs about their ability to overcome fatigue, and the scheduling of daily activities, with an aim to increase physical activities in daily life and finally reduce the level of fatigue.
  Each participant will meet a therapist in six face-to-face sessions. Each session will be about one hour and be two weeks apart. During the sessions, the participant will discuss with the therapist their problems related to fatigue and work through an intervention manual to learn skills to overcome these problems.
  Interventions: Behavioral: A brief psychological intervention

INTERVENTIONS:
Behavioral: A brief psychological intervention — This intervention is based on the principle of cognitive-behavioral therapy

SUMMARY:
Stroke is a leading cause of adult disability in the community. Fatigue affects about a third of stroke survivors. It results in difficulty taking part in everyday activities, and increases risk of hospitalization and death after stroke. Despite of its high prevalence and distressing consequences, there is no effective treatment.

Psychological interventions have improved fatigue in patients with other conditions such as multiple sclerosis. These interventions primarily target patients' beliefs about overcoming fatigue and their physical activities in daily life. Also studies indicated that post-stroke fatigue is associated with mood. Based on this knowledge, the investigator has designed a brief psychological intervention for post-stroke fatigue.

The current study is a feasibility study to test the adequacy of intervention manuals and the feasibility of trial processes. This study will need 12 stroke survivors who have post-stroke fatigue and are over three months but within two years after their stroke. Stroke survivors with severe depression or having insufficient capability in cognition or communication will not be included. The investigator will check their eligibility by questionnaires and interviews and then invite eligible people to take part in the study.

This intervention will be delivered by a therapist (a clinical psychologist) to each participant through six face-to-face therapy sessions. Each session will be about one hour and be two weeks' apart. During the sessions, participants will discuss with the therapist their fatigue problems, and, with the support from the therapist, work out ways to solve their problems. One month after the last face-to-face session, each participant will receive a feedback session by telephone from the therapist. Each participant will be followed up to three months after the last face-to-face session.

After all participants complete their feedback sessions, the investigator will invite them to a group meeting to share their experiences of taking part in this trial and makes suggestions as how their experiences of this intervention, and also of this trial, could be improved.

DETAILED DESCRIPTION:
This is a feasibility study to test a brief psychological intervention for post-stroke fatigue. 12 stroke survivors with post-stroke fatigue will be recruited for this study. This intervention has been adapted from similar interventions that have improved fatigue in other conditions, such as multiple sclerosis, cancer and chronic fatigue syndrome. Like in other conditions, fatigue in stroke survivors is associated with low mood, people's beliefs about overcoming fatigue, and reduced physical activity. This intervention will target patients' mood, their beliefs about their ability to overcome fatigue, and the scheduling of daily activities, with an aim to increase physical activities in daily life and finally reduce the level of fatigue.

Following the relevant guideline of the United Kingdom (UK) Medical Research Council, the investigators will perform a sequence of trials to test the feasibility, safety and effectiveness of this intervention. Current study is an initial stage to test the feasibility of the intervention, i.e. whether this brief psychological intervention could be adequately delivered to people with post-stroke fatigue on an individual basis. To standardize the therapeutic components of this psychological intervention, this intervention will be delivered by a clinical psychologist in the current study. In subsequent trials, the intervention will then be adapted to be delivered by stroke nurses, which is a more practical situation within the National Health Service of the United Kingdom.

Check for eligibility and consent for participation: the investigator will send mails to stroke survivors who had a stroke between the past three to 24 months to invite them to take part in a survey for post-stroke fatigue and depression. For those who have post-stroke fatigue and do not have severe depression, they will be invited to a face-to-face meeting with the investigator. At this meeting, the investigator will further check the eligibility of each potential participant and answer his/her questions about this study. If the potential participant is willing to take part in the trial, him/her will be asked to sign a consent form for participation.

Baseline assessment of clinical outcomes: after signing the consent, the participant will be asked to complete four questionnaires for baseline assessment:

1. Fatigue Assessment Scale
2. Case definition of post-stroke fatigue
3. Nottingham Extended Activities of Daily Living
4. Stroke Impact Scale

Therapy sessions: each participant will be attending six face-to-face sessions over a period of eleven weeks in the hospital. Each session will last for about one hour, where the participant will meet a therapist (a clinical psychologist) of this intervention. With the support from the therapist, the participant will work through an intervention manual to learn skills to overcome their problems related to fatigue, especially for physical activity, mood and sleep. There will be intervals of two weeks between sessions. During the intervals, the participant will be asked to keep a diary to record their daily activities and sleep, to put into action things they have agreed with the therapist (including doing more activity), or to read sections of the intervention manual.

Post-treatment assessment of clinical outcomes: participants will three assessments of clinical outcomes, i.e. immediately after completing all six treatment sessions, one month after treatment, and three-month after treatment.

1. Fatigue (Fatigue Assessment Scale and a case definition of post-stroke fatigue)
2. Depression (Patient Health Questionnaire-9)
3. Independence in daily life (Nottingham Extended Activities of Daily Living)
4. Health-related quality of life (Stroke Impact Scale)

An interim analysis will be performed after one-month assessment and the final analysis will be performed after the three-month assessment. Before- and after- treatment assessments will show whether the intervention is beneficial for the above aspects and whether these benefits could be maintained. The investigator will then write to each participant to inform them of the individual results of both analyses.

Feedback session: at the time of one-month assessment, the participant will be asked to fill a feedback form for their experience of this intervention and the trial. The investigator will analyze the results of this feedback form as well as the results of one-month assessment, and then inform both the participant and the therapist of the individual results. Then the therapist will carry out a feedback session with each participant by telephone (about one hour). During this session, they will discuss the results of assessments and any difficulties that the participant may have experienced in the past month. They will also agree a plan to make further improvement.

Fatigue is a chronic symptom which would require a long term for recovery. Thus this intervention with six treatment sessions is expected to be an intensive initial program for the recovery of post-stroke fatigue, from which participants will learn skills to overcome fatigue-related problems that they can use in daily life. Thus the therapist will encourage participants to continue using these skills in their daily life even after completing the therapy sessions.

Feedback meeting: after all participants have completed their feedback sessions, the investigator will invite them to a feedback meeting. This meeting will be facilitated by the Chief Investigator of this study. At this meeting, participants will share their experience in taking part in this trial, discuss any difficulties they have experienced, and make suggestions to improve this intervention and the trial processes.

ELIGIBILITY:
Inclusion Criteria:

* Had a clinical diagnosis of stroke in the past three to 24 months (including minor stroke)
* Have post-stroke fatigue
* Over 18 years old
* Live in the Lothian area, Scotland

Exclusion Criteria:

* Have severe depression (with a total score of the Patient Health Questionnaire-9 of 15 or more)
* Have severe cognitive deficits
* Have severe aphasia
* Have significant difficulty in verbal communication
* Medically unstable or have another unfavorable condition that could impact results (e.g. substance abuse)
* Being in the nursing home
* Currently in another research study that might affect fatigue or add significant burden to participants, e.g. studies have outcome measures for fatigue or involve physical training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simiao Wu, MD, PhD, Principal Investigator — Centre for Clinical Brain Sciences, University of Edinburgh, United Kingdom
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Background] Wu S, Barugh A, Macleod M, Mead G. Psychological associations of poststroke fatigue: a systematic review and meta-analysis. Stroke. 2014 Jun;45(6):1778-83. doi: 10.1161/STROKEAHA.113.004584. Epub 2014 Apr 29. PMID 24781083
- [Background] Duncan F, Wu S, Mead GE. Frequency and natural history of fatigue after stroke: a systematic review of longitudinal studies. J Psychosom Res. 2012 Jul;73(1):18-27. doi: 10.1016/j.jpsychores.2012.04.001. Epub 2012 Apr 29. PMID 22691555
- [Background] Wu S, Mead G, Macleod M, Chalder T. Model of understanding fatigue after stroke. Stroke. 2015 Mar;46(3):893-8. doi: 10.1161/STROKEAHA.114.006647. Epub 2015 Feb 3. No abstract available. PMID 25649798
- [Result] Wu S, Chalder T, Anderson KE, Gillespie D, Macleod MR, Mead GE. Development of a psychological intervention for fatigue after stroke. PLoS One. 2017 Aug 17;12(8):e0183286. doi: 10.1371/journal.pone.0183286. eCollection 2017. PMID 28817725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was started in July 2014 and completed in October 2014. Participants were recruited through three approaches, including patients discharged from the Stroke Ward, patients visiting the Stroke Clinic, and those visited by the stroke nurses in the community.
Groups:
- Psychological Intervention: All participants were enrolled in this group, receiving a psychological intervention for the treatment of post-stroke fatigue.
Period: Overall Study
Arm/Group | Psychological Intervention
Started | 12
Completed | 8
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Other health conditions | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Baseline characteristics of eight participants who completed all treatment sessions
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8
Fatigue Assessment Scale [Mean (Standard Deviation); unit: units on a scale] — The total score of FAS ranges from 10 to 50, with higher scores indicating worse outcomes.
  units on a scale | 26.5 (8.0)
Case definition of post-stroke fatigue [Number; unit: participants] — To fulfill this case definition, the patient should describe feelings of tiredness, lack of energy or fatigue or increased need to rest as opposed to lack of motivation or boredom. Also the patient should have felt fatigue everyday or nearly everyday for at least 2 weeks in the past month. Finally, fatigue must be perceived as a problem and affect everyday activities.
  participants
    Fulfilling case definition | 5
    Not fulfilling case definition | 3
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — The total score of PHQ-9 ranges from 0 to 27, with higher scores indicating worse outcomes.
  units on a scale | 7.6 (4.3)
Nottingham Extended Activities of Daily Living [Mean (Standard Deviation); unit: units on a scale] — The total score of NEADL ranges from 0 to 22, with higher scores indicating better outcomes
  units on a scale | 20.8 (0.9)
Stroke Impact Scale - General rating of recovery [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, presenting the percentage of recovery from stroke.
  units on a scale | 74.8 (16.7)
Stroke Impact Scale - Physical Strength [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 89.06 (9.88)
Stroke Impact Scale - Memory and Thinking [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 75.45 (21.29)
Stroke Impact Scale - Emotion [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 65.97 (26.13)
Stroke Impact Scale - Communication [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 80.36 (23.30)
Stroke Impact Scale - Daily Activities [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 93.44 (6.54)
Stroke Impact Scale - Mobility [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 87.50 (15.14)
Stroke Impact Scale - Hand Function [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 93.75 (9.54)
Stroke Impact Scale - Social Activity [Mean (Standard Deviation); unit: units on a scale] — The score ranges from 0 to 100, with higher scores indicating better outcomes.
  units on a scale | 67.85 (24.55)

OUTCOME MEASURES:

1. Secondary Outcome: Fatigue Assessment Scale (FAS)
Description: This is the primary clinical outcome for this intervention (but clinical outcomes are all secondary outcomes for this pilot feasibility study).
  The total FAS score ranges from 10 to 50, with higher scores indicating worse outcomes of fatigue severity.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: Eight participants who completed all treatment sessions were included for data analysis
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 17.25 (8.56)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in fatigue scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.03, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 9.250, 95% CI 2-sided [1.398 to 17.102], Standard Error of Mean 3.321 — P values below 0.05 are considered statistically significant in this study

2. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The total PHQ-9 score ranges from 0 to 27, with higher scores indicating worse outcomes of depressive symptoms.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 5.00 (6.32)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in depression scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.10, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 2.625, 95% CI 2-sided [-0.687 to 5.937], Standard Error of Mean 1.401 — P values below 0.05 are considered statistically significant in this study

3. Secondary Outcome: Nottingham Extended Activities of Daily Living (NEADL)
Description: The total NEADL score ranges from 0 to 22, with higher scores indicating better outcomes of independence.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 21.00 (1.07)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in independence scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.45, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.250, 95% CI 2-sided [-0.991 to 0.491], Standard Error of Mean 0.313 — P values below 0.05 are considered statistically significant in this study

4. Secondary Outcome: Stroke Impact Scale (SIS) - General Rating of Recovery
Description: The general rating scale on the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes of recovery.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 88.63 (15.16)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in scores of general rating of recovery between baseline and three-month assessments; Test type: Superiority or Other; p = 0.03, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -13.875, 95% CI 2-sided [-25.769 to -1.981], Standard Error of Mean 5.030 — P values below 0.05 are considered statistically significant in this study

5. Secondary Outcome: SIS - Physical Strength
Description: The physical strength subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 89.84 (12.47)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in physical strength scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.89, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.781, 95% CI 2-sided [-14.010 to 12.448], Standard Error of Mean 5.594 — P values below 0.05 are considered statistically significant in this study

6. Secondary Outcome: SIS - Memory and Thinking
Description: The memory and thinking subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 87.05 (18.00)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in memory and thinking scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -2.105, 95% CI 2-sided [-7.729 to 3.519], Standard Error of Mean 2.378 — P values below 0.05 are considered statistically significant in this study

7. Secondary Outcome: SIS - Emotion
Description: The emotion subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 84.38 (18.84)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in emotion scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -18.403, 95% CI 2-sided [-30.624 to -6.183], Standard Error of Mean 5.168 — P values below 0.05 are considered statistically significant in this study

8. Secondary Outcome: SIS - Communication
Description: The communication subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 87.50 (17.91)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in communication scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.10, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -7.142, 95% CI 2-sided [-15.883 to 1.598], Standard Error of Mean 3.696 — P values below 0.05 are considered statistically significant in this study

9. Secondary Outcome: SIS - Daily Activities
Description: The daily activities subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 95.94 (5.33)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in daily activities scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.09, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -2.500, 95% CI 2-sided [-5.455 to 0.455], Standard Error of Mean 1.250 — P values below 0.05 are considered statistically significant in this study

10. Secondary Outcome: SIS - Mobility
Description: The mobility subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 91.32 (13.96)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in mobility scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.03, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -3.821, 95% CI 2-sided [-7.091 to -0.551], Standard Error of Mean 1.382 — P values below 0.05 are considered statistically significant in this study

11. Secondary Outcome: SIS - Hand Function
Description: The hand function subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 95.63 (8.63)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in hand function scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.58, t-test, 2 sided — The critical level was adjusted for the multiple comparisons for the eight subscales of the Stroke Impact Scale; Paired t-test; Mean Difference (Final Values) = -1.875, 95% CI 2-sided [-9.594 to 5.844], Standard Error of Mean 3.264 — P values below 0.05 are considered statistically significant in this study

12. Secondary Outcome: SIS - Social Activity
Description: The social activity subscale of the Stroke Impact Scale 3.0, of which the score ranges from 0 to 100, with higher scores indicating better outcomes.
Time Frame: 3 months after the end of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
units on a scale | 82.42 (19.90)
Statistical Analysis 1: Comparison: Intervention Group; Null hypothesis: there was no difference in social activity scores between baseline and three-month assessments; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — The critical level was adjusted for the multiple comparisons for the eight subscales of the Stroke Impact Scale; Paired t-test; Mean Difference (Final Values) = -14.576, 95% CI 2-sided [-23.304 to -5.847], Standard Error of Mean 3.691 — P values below 0.05 are considered statistically significant in this study

13. Primary Outcome: Feasibility of Recruitment Process
Description: The numbers of stroke patients involved at each stage of recruitment were reported under this outcome.
Time Frame: 3 months after the end of treatment
Measure: Number; unit: participants
Groups:
- Intervention Group: This outcome presents the recruitment process. However, only eight participants who completed all treatment sessions were included for further analysis of clinical outcomes.
Arm/Group | Intervention Group
Number analyzed (Participants) | 120
participants
  Initially approached patients | 120
  Responding patients | 49
  Eligible patients | 20
  Consented patients | 12

14. Primary Outcome: Attendance of Treatment Sessions
Description: Number of participants who completed all treatment sessions.
Time Frame: 3 months after the end of treatment
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
participants | 8

15. Primary Outcome: Feasibility of Telephone-delivered Booster Sessions
Description: Numbers of participants who attended the booster session as planned and those who rearranged the session
Time Frame: 3 months after the end of treatment
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
participants
  Attended as planned | 1
  Rearranged | 7

16. Primary Outcome: Feasibility of Follow-up Assessment at Three Months After the End of Treatment
Description: Numbers of participants who completed and returned the questionnaires on time (as required) and of those who delayed the completion.
Time Frame: 3 months after the end of treatment
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
participants
  On time | 6
  Delayed | 2

ADVERSE EVENTS:
Time Frame: From the beginning to the end of treatment (11 weeks).
Arm/Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
The aim of this single-arm pilot study was to test the feasibility of the intervention programme. This study can not inform the sample size calculation or efficacy of the intervention, which should be investigated in randomised controlled trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No